CLINICAL TRIAL: NCT02088931
Title: A Pilot Trial of CD4+CD127lo/-CD25+ Polyclonal Treg Adoptive Immunotherapy in Renal Transplant Recipients
Brief Title: Treg Adoptive Therapy for Subclinical Inflammation in Kidney Transplantation
Acronym: TASK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSFTX412ST
Record Dates: First submitted 2014-01-13; First posted 2014-03-17 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Late Complication From Kidney Transplant
Keywords: Tregs; Kidney transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single infusion polyclonal Treg (Experimental): 3 subjects with inflammation on their 6-month surveillance biopsy following renal transplantation will receive a single infusion of a target of 320 million ex vivo selected and expanded autologous polyclonal Tregs.
  After the therapy visit the patient will return for a total of nine (9) more visits for the main part of the study: 1 and 4 days after therapy, then once a week for 4 weeks, and then 3, 6, and 12 months after you get the therapy.
  Interventions: Biological: Treg infusion

INTERVENTIONS:
Biological: Treg infusion — At the time of Treg infusion (day 0), maintenance immunosuppression will remain unchanged which consists of TAC, MPA and steroids. On follow-up biopsy 2 weeks after Treg infusion, the inflammatory load will be assessed by computer assisted image analysis looking at the number of infiltrating cells per square mm as well as the percentage of renal cortex infiltrated with lymphocytes. If the inflammatory load has decreased by ≥50% and infused Tregs are observed in the allograft, everolimus will be started at 1.5 mg bid and the dose of tacrolimus will be decreased by 50%. After 2 weeks, tacrolimus will be discontinued. These patients will remain on everolimus, mycophenolic acid and prednisone through the end of the study and the follow-up period. If on the 2-week follow-up biopsy, there is no decrease in the inflammatory load or there is a decrease <50%, no change will be made to the maintenance immunosuppressive regimen consisting of TAC, MPA and prednisone.

SUMMARY:
The purpose of this study is to test the safety of the experimental therapy of a single infusion of Regulatory T cells (Tregs). The investigators want to find out what effects, good or bad, Tregs will have on the kidney transplant patients.

There are different types of T cells. This study uses Regulatory T cells (Tregs), which are found in the blood and are part of the immune system that stops other immune cells from working. Tregs help to turn off the immune system after other immune cells have finished tackling outside infections, and Tregs keep the immune system in check so that the body does not attack itself. The researchers are hoping that, by giving an infusion of Tregs that the attack on the kidney can be stopped and kidney function will be stabilized. It is not known if the Treg experimental therapy can stop the inflammation in the kidney.

In this study, the researchers will take some of Tregs from the patient, multiply them in the laboratory, and then infuse them back into the patient. The procedure used to multiply Tregs is an experimental process performed in the laboratory. Similar procedures done with mice have been shown to reverse inflammation but it is not known whether the results will be the same in humans. This therapy has not yet been done in humans outside of a research study.

DETAILED DESCRIPTION:
This is an open-label single dose pilot study in which 3 subjects with inflammation on their 6-month surveillance biopsy following renal transplantation will receive a single infusion of a target of 320 million cells ex vivo selected and expanded autologous polyclonal Tregs.

AAt the time of Treg infusion (day 0), the immnosuppression will remain unchanged and consists of tacrolimus and mycophenolate acid with or without steroids. On the follow up biopsy, 2 weeks after the Treg infusion, the inflammatory load will be assessed by computer assisted image analysis looking at thenumber of infiltrating cells per square mm as well as the percentage of renal cortex infiltrated with lymphocytes. If the inflammatory load has decreased by ≥50% and infused Tregs are observed in the allograft, everolimus will be started at 1.5 mg bid and the dose of tacrolimus will be decreased by 50%. After 2 weeks, tacrolimus will be discontinued. These patients will remain on everolimus and mycophenolic acid with or without prednisone through the end of the study and the follow up period. If on the 2-week follow-up biopsy, there is no decrease in the inflammatory load or there is a decrease <50%, no change will be made to the maintenance immunosuppressive regimen consisting of tacrolimus, mycophenolic acid with or without prednisone. immunosuppression. All prescribing physicians are enrolled in and will participate in the FDA Mycophenolate Risk Evaluation and Mitigation Strategy.

Subjects will be enrolled at 4-6 week intervals. The first subject will receive an infusion and will be observed for 3 weeks prior to treatment of the remaining subjects. The study team (IND sponsor, protocol chair, and medical monitor) and the members of the DSMB will review the safety data of the first subject prior to proceeding.

If no grade 3 or higher related adverse event is observed, subsequent subjects may be treated. Otherwise treatment will be suspended pending review.

ELIGIBILITY:
Inclusion Criteria:

1. Recipients of primary renal transplants age 18-65 years with no donor specific antibodies prior to transplantation
2. Stable renal function (cGFR), no history of acute rejection and proteinuria less than 500 mg/24 hours.
3. Maintenance immunosuppression consisting of tacrolimus and mycophenolate mofetil/mycophenolic acid with or without prednisone
4. Protocol renal allograft biopsy at 6 months with findings of 5%-25% inflammation (Banff t0 or t1)without evidence of rejection (Banff t0 or t1<5%)
5. Blood PCR for BK less than 1000 copies/ml, and urine less than 500,000 copies/ml
6. History of positive EBV serology
7. Current immunizations including TdAP, hepatitis B, pneumococcal and seasonal influenza vaccines

Exclusion Criteria:

1. Recipients of 6-antigen HLA matched kidney transplants from living or deceased donors
2. Subjects with history of prior kidney transplant
3. History of transplant renal artery stenosis
4. History of wound healing complication following transplant surgery
5. Known hypersensitivity to tacrolimus, mycophenolate mofetil/mycophenolic acid, or everolimus
6. Subjects with history of autoimmune disease
7. Hematocrit < 33%; leukocytes <3,000/μL; neutrophils <1,500/μL; lymphocytes <800/μL; platelets <100,000/μL
8. Any current active infection
9. Serologic evidence of HIV-1 or HIV-2 infection
10. Evidence of current hepatitis B as demonstrated by HBsAg or circulating hepatitis B genomes
11. Serologic evidence of hepatitis C infection
12. Detectable circulating CMV genomes or active infection or high risk for CMV (CMV seronegative recipient receiving a kidney from a CMV seropositive donor)
13. Detectable circulating EBV genomes
14. History of positive PPD skin test, which was untreated.
15. Subjects who may potentially require live virus vaccines within the first 12 months of the study
16. History of malignancy (including squamous cell carcinoma of the skin or cervix) except adequately treated basal cell carcinoma
17. Any chronic illness or prior treatment which in the opinion of the investigator should preclude participation in the trial
18. Pregnant or breastfeeding women, any female who is unwilling to use a reliable and effective form of contraception for 2 years after Treg dosing, and any male who is unwilling to use a reliable and effective form of contraception for 3 months after Treg dosing
19. Tregs present in peripheral blood at less than 30/µL

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2014-03; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Adverse Events. | 1 year
  Participants will be assessed for adverse events on days 0-1 (Treg infusion) and on days 4,7,14,21,28,84,180, and 360 (1 year).
Patient Survival | 3 years
  Patient survival at 1 year and 3 years post renal transplantation.
Renal Allograft Survival | 3 years
  Renal allograft survival at 1 year and 3 years post renal transplantation.
Renal Allograft Dysfunction | 1 year
  Incidence of renal allograft dysfunction during the 1 year follow-up period post Treg infusion.

SECONDARY OUTCOMES:
Presence of Intragraft Tregs in the Renal Allograft Biopsy | 2 weeks
  Treg infiltration will be measured in the renal allograft on the post infusion kidney biopsy to observe the persistence of deuterium-labeled Tregs within the allograft.
Change in circulating Treg Cells | 2 weeks
  Percentage of circulating Treg cells detected using deuterium labeling in the allograft biopsy.

OTHER OUTCOMES:
Change from Baseline in Urinary Protein | 1 year
  Assess surrogate markers of immune response by measuring changes in urinary protein and reflecting immune infiltration, inflammation, and tubular injury. (composite measure)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Vincenti, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Nankivell BJ, Borrows RJ, Fung CL, O'Connell PJ, Allen RD, Chapman JR. Natural history, risk factors, and impact of subclinical rejection in kidney transplantation. Transplantation. 2004 Jul 27;78(2):242-9. doi: 10.1097/01.tp.0000128167.60172.cc. PMID 15280685
- [Result] Kee TY, Chapman JR, O'Connell PJ, Fung CL, Allen RD, Kable K, Vitalone MJ, Nankivell BJ. Treatment of subclinical rejection diagnosed by protocol biopsy of kidney transplants. Transplantation. 2006 Jul 15;82(1):36-42. doi: 10.1097/01.tp.0000225783.86950.c2. PMID 16861939
- [Result] Sakaguchi S, Yamaguchi T, Nomura T, Ono M. Regulatory T cells and immune tolerance. Cell. 2008 May 30;133(5):775-87. doi: 10.1016/j.cell.2008.05.009. PMID 18510923
- [Result] Tang Q, Bluestone JA, Kang SM. CD4(+)Foxp3(+) regulatory T cell therapy in transplantation. J Mol Cell Biol. 2012 Feb;4(1):11-21. doi: 10.1093/jmcb/mjr047. Epub 2011 Dec 14. PMID 22170955